CLINICAL TRIAL: NCT06361251
Title: Interventional, Monocentric, Double-blind Randomized Category 2b Study Evaluating the Evaluation of the Tolerance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots (Solar and Senile Lentigines, Post -Inflammatory Hyperpigmentation (Pih)) on the Face
Acronym: CS5_10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_10
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lentigo; Solar Lentigo; Post Inflammatory Hyperpigmentation
Keywords: cryotherapy; brown spots
MeSH Terms: conditions — Lentigo; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Proof of concept study concerning 2 prototypes of cyto-selective cryotherapy devices corresponding to a modified CE marked medical device (ref: 822-v1).
Who Masked: Participant, Investigator
Masking Description: Double blind (participant and care provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (EC14_4osc) (Experimental): (EC14_4osc) 1 application every week for a total of 6 applications
  Interventions: Device: CRYONOVE (EC14_4osc)
- (EC-05_1osc) (Experimental): (EC-05_1osc) 1 application every two weeks for a total of 6 applications
  Interventions: Device: CRYONOVE (EC05osc)

INTERVENTIONS:
Device: CRYONOVE (EC14_4osc) — The prototype is a variant version from that of a CE marked MD already commercialized (Cryobeauty mains, Cryobeauty Pharma SAS, France) which produces a cryogenic spray sequence (EC14). The prototype is intended to treat pigmented spots of the face (PIH spots and senile and solar lentigos).
  Arms: (EC14_4osc)
Device: CRYONOVE (EC05osc) — The prototype is a variant version from that of a CE marked MD already commercialized (Cryobeauty mains, Cryobeauty Pharma SAS, France) which produces a cryogenic spray sequence (EC05). The prototype is intended to treat pigmented spots of the face (PIH spots and senile and solar lentigos).
  Arms: (EC-05_1osc)

SUMMARY:
The goal of this clinical trial is to compare the 2 different prototype of cytoselectivecryotherapy devices (name of the devices : CRYONOVE) use in brown spots on the face of subject from different ethnicities. The main questions it aims to answer are:

* the tolerance of 2 prototypes of cyto-selective cryotherapy treatments
* the performance of 2 prototypes of cyto-selective cryotherapy treatments Participants will be treated for each spots with a definied prototype during 6 treatment visits.

Researchers will compare the tolerance and performance of the 3 prototypes.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed a written informed consent form (ICF) to participate in the investigation obtained according to ISO 14155:2020 - Good Clinical Practice (GCP);
2. Healthy male and female participants, 18 to 75 years old (inclusive), and Fitzpatrick's skin type (V-VI);
3. Melanin-rich ethnicity skins;
4. Presenting at least two brown spots on the face with ≥ 3 and ≤ 6 mm in diameter;
5. Female of non-childbearing potential, defined as woman without uterus and/or both ovaries, surgically sterile (at least 6 months prior to Screening visit) or post-menopausal (at least one year post cessation of menses);
6. Female of childbearing potential who has been, in the opinion of the Investigator, using an approved method of birth control for at least 1 month prior to Screening visit and agreeing to continue adequate contraception during the entire study period;

   Reliable methods of contraception are:
   * hormonal methods or intrauterine device in use since at least 1 month prior to Screening visit and during the investigation period;
   * bilateral tubal ligation since at least 3 months prior to Screening visit and during the investigation period;
   * barrier methods in use at least 14 days prior to Screening visit;
   * vasectomized partner;
   * sexual abstinence defined as refraining from heterosexual intercourse for at least 3 months prior to Screening visit and during the entire period of risk associated with the study products.
7. Participant who has not been exposed to UV within at least two months prior to the screening visit and agreeing to avoid exposure to UV radiation (tanning beds, phototherapy and sunlight) for the whole study duration. A sun-protection cream will be distributed to the participants to use in case of sun exposure;
8. Having undergone a general clinical examination attesting to his/her ability to participate in the study.
9. Participant able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on Investigator's judgement;
10. No suspicion of carcinoma after investigation by a dermatologist

Exclusion Criteria:

1. Female participant who is pregnant, parturient or breast feeding;
2. Female participant of childbearing potential having a positive urinary pregnancy test at Day 0;
3. Having performed cosmetic treatments (e.g., exfoliants, scrubs or self-tanners, facial UV) in the month before the start of the study on the face (see restrictions paragraph);
4. Having performed cosmetic or aesthetic treatments by a dermatologist (e.g., laser, IPL, peeling, creams, cryotherapy) in the last 6 months on the face;
5. Receiving systemic or local treatment (e.g., dermocorticoids, corticosteroids, diuretics) likely to interfere with the evaluation of the parameter studied;
6. Person affected by dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (e.g., people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome);
7. Person with clinically significant skin condition on the tested area (e.g., active eczema, psoriasis, rosacea, scleroderma, acne, dermatitis) or presence on the tested area of skin lesions, scars, tattoos;
8. Concomitant participation in other clinical trials/investigations or participation in the evaluation of any IMD/IP during 2 months before this study;
9. Unable to follow the requirements of the protocol.Vulnerable: whose ability or freedom to give or refuse consent is limited.
10. Major protected by law (tutorship, curatorship, safeguarding justice...).
11. Unable to be contacted urgently over the phone.
12. Unable to communicate or cooperate with the Investigator due to poor mental development, language problems (unable to read and write English language) or impaired cerebral function;
13. Currently participating in another clinical study or being in an exclusion period of another clinical study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Tolerance | [Time Frame: Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70]
  Evaluate the evolution of the scores given by the dermatologist or the participant on the following items :
  Hyperpigmentation (IGA scale)* Hypopigmentation Erythema, oedema, micro-bruise, hematoma, dryness, desquamation, fissures / cracks, roughness, crust Skin sensation (tightness, stinging, itching, warm and burning sensations) Day 0: Pain after each treatment (5 min. rest between two treatments) Other unexpected events
  *: IGA Scale : Investigator's Global Assessment - Scale in 6 points (0 to 5) 0 = clear of hyperpigmentation
  1. = almost clear of hyperpigmentation
  2. = mild, but noticeable hyperpigmentation
  3. = moderate hyperpigmentation (medium brown in quality)
  4. = severe hyperpigmentation (dark brown in quality)
  5. = very severe hyperpigmentation (very dark brown, almost black in quality)

SECONDARY OUTCOMES:
Performance (Acquisitions C-cube) | [Time Frame: Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70]
  --> Performance assesment :
  • Standardized photographs will be taken before the treatment at each visit (C-Cube acquisition without analysis) - illustration only

CONTACTS AND LOCATIONS:
Overall Officials: Victoria DAUPHANT, Study Chair — Dermatech
Locations (1):
- SMU - Photobiology Laboratory, Sefako Makgatho Health Sciences University, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: No